CLINICAL TRIAL: NCT01358968
Title: A Study in Cancer Patients to Evaluate the Ability of LY2603618 to Act as an Inhibitor of CYP2D6 Using Desipramine as a Probe Substrate
Brief Title: A Drug Interaction Study to Assess the Effect of LY2603618 on the Metabolic Pathway of Desipramine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13526; I2I-MC-JMMI (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-05-20; First posted 2011-05-24 (Estimated); Results first posted 2018-10-25 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-03

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — LY2603618; Desipramine; Pemetrexed; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY2603618 (Experimental): Single 50 milligrams (mg) oral dose of desipramine on day 1 of study period 1. Single 275 mg intravenous infusion over one hour of LY2603618 followed by single 50 mg oral dose of desipramine on day 1 of study period 2. Participants may then receive additional doses of LY2603618 in combination as follows: 1000 milligrams per square meter (mg/m²) intravenous administration over 30 minutes of gemcitabine on days 1, 8 and 15 and 230 mg intravenous dose of LY2603618 on days 2, 9 and 16 of 28-day cycles OR 500 mg/m² intravenous administration over 10 minutes of pemetrexed on day 1 and 275 mg intravenous dose of LY2603618 on day 2 of 21-day cycles.
  Participants will be allowed to continue to receive the combination therapy until fulfilling one of the criteria for discontinuation, such as unacceptable toxicity or disease progression.
  Interventions: Drug: LY2603618; Drug: Desipramine; Drug: Pemetrexed; Drug: Gemcitabine

INTERVENTIONS:
Drug: LY2603618 — Administered intravenously as a 1-hour infusion.
Drug: Desipramine — Administered orally
Drug: Pemetrexed — Administered intravenously as a 10-minute infusion.
  Other Names: ALIMTA®; LY231514
Drug: Gemcitabine — Administered intravenously as a 30-minute infusion.
  Other Names: Gemzar®; LY188011

SUMMARY:
The purpose of this study is to assess the effect LY2603618 on a protein [enzyme cytochrome P (CYP) 2D6] which is involved in the metabolic pathway of Desipramine in participants with cancer. This is a drug interaction study so the treatment of the disease will not be the main purpose of the study.

The study involves two single doses of 50 milligrams (mg), 1 tablet by mouth, on Day 1 of Period 1 and 2. In Period 1 Desipramine will be administered alone. In Period 2 Desipramine will be administered in combination with LY2603618. LY2603618 will be administered as a 275mg intravenous (IV) infusion over 1 hour (hr).

Desipramine will be administered at the end of the LY2603618 infusion. Information about any side effects that may occur will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Have a histological or cytological diagnosis of cancer (solid tumor), with clinical or radiologic evidence of locally advanced and/or metastatic disease, for which no life-prolonging therapy exists (that is, refractory to standard therapy and/or therapies known to provide clinical benefit, or for which no standard therapy exists). Note: Participants who have had progressive disease after receiving pemetrexed for metastatic disease are excluded from receiving the combination with pemetrexed during the safety extension study. Participants who have had progressive disease after receiving gemcitabine for metastatic disease are excluded from receiving the combination with gemcitabine during the safety extension study.
* Have a body surface area (BSA) greater than or equal to 1.37 square meters (m²)
* Have given written informed consent prior to any study-specific procedures
* Have adequate hematologic, hepatic and renal function
* Have a performance status of less than or equal to 2 on the Eastern Cooperative Oncology Group (ECOG) scale
* Have discontinued all previous treatments for cancer, including chemotherapy, radiotherapy, anticancer hormone therapy or other investigational therapy for at least 30 days prior to study entry and recovered from the acute effects of therapy (at least 42 days for mitomycin-C or nitrosoureas, or 60 days for biologics)
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* Males and females with reproductive potential: Must agree to use medically approved contraceptive precautions during the study and for at least 3 months following the last dose of study drug
* Females with childbearing potential: Have had a negative serum pregnancy test less than or equal to 7 days before the first dose of study drug and must also not be breastfeeding
* Have an estimated life expectancy, in the judgment of the investigator, that will permit the participant to complete 1 full cycle of treatment beyond the drug interaction portion of the study (approximately 8 weeks)
* Are able to swallow tablets
* Prior radiation therapy for treatment of cancer is allowed to <25% of the bone marrow and participants must have recovered from the acute toxic effects of their treatment prior to study enrollment. Prior radiation to the whole pelvis is not allowed. Prior radiotherapy must be completed at least 4 weeks before study entry.

Exclusion Criteria:

* Have received treatment within 28 days of the initial dose of study drug with an experimental agent for noncancer indications that has not received regulatory approval for any indication
* Poor metabolizer (PM) status for CYP2D6 (genotyped)
* Have previously completed or withdrawn from this study or any other study investigating LY2603618 or any other checkpoint kinase one (Chk1) inhibitor
* Have known allergy to gemcitabine, pemetrexed, desipramine or LY2603618 or any ingredient of gemcitabine, pemetrexed, desipramine or LY2603618 (like Captisol®)
* Have serious preexisting medical conditions (left to the discretion of the investigator) other than advanced cancer
* Have symptomatic central nervous system (CNS) malignancy or metastasis (screening not required). Participants with treated CNS metastases are eligible for this study if they are not currently receiving corticosteroids and/or anticonvulsants, and their disease is asymptomatic and radiographically stable for at least 90 days.
* Have current hematologic malignancies or either acute or chronic leukemia
* Have an active fungal, bacterial, and/or known viral infection including human immunodeficiency virus (HIV) or viral (A, B, or C) hepatitis (screening is not required)
* Have QTc interval of >500 milliseconds (msec) on screening electrocardiogram (ECG)
* Have ECG abnormalities on the screening ECG such as significant conduction abnormalities, ischemic changes (such as prior Q-wave myocardial infarction and/or marked ischemic ST- and T-wave), arrhythmias (such as persistent or paroxysmal ventricular or supraventricular arrhythmias, including atrial fibrillation), or other ECG abnormalities that would put the participant at unnecessary risk in the opinion of the investigator
* Drugs with narrow therapeutic windows and that are also known substrates of CYP2D6 or drugs that are classified as sensitive substrates of CYP2D6 are excluded
* Drugs or herbal supplements that are known inhibitors of CYP2D6 are excluded during the study, and during the 30-day period (or a minimum of 5 half-lives, whichever is less) prior to study start
* Participants who have an average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females), or participants unwilling to stop alcohol consumption for 24 hours before the study through the end of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-06; Primary Completion 2012-04 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-371-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a nonrandomized, open-label, fixed-sequence, 2-period study followed by a continued access phase.
Groups:
- Desipramine (Period 1): Single 50-milligram (mg) oral dose of desipramine on Day 1 of Study Period 1.
- LY2603618 + Desipramine (Period 2): Single 275-mg intravenous infusion over one hour of LY2603618 followed by single 50-mg oral dose of desipramine on Day 1 of Study Period 2.
- LY2603618 + Gemcitabine (Continued Access): 1000-milligrams per square meter (mg/m²) intravenous administration over 30 minutes of gemcitabine on Days 1, 8 and 15 and 230-mg intravenous infusion over one hour of LY2603618 on Days 2, 9 and 16 of 28-day cycles during continued access phase.
  Participants were allowed to continue to receive the combination therapy until fulfilling one of the criteria for discontinuation, such as unacceptable toxicity or disease progression.
- LY2603618 + Pemetrexed (Continued Access): 500-mg/m² intravenous administration over 10 minutes of pemetrexed on Day 1 and 275-mg intravenous infusion over one hour of LY2603618 on Day 2 of 21-day cycles during continued access phase.
  Participants were allowed to continue to receive the combination therapy until fulfilling one of the criteria for discontinuation, such as unacceptable toxicity or disease progression.
Period: Period 1
Arm/Group | Desipramine (Period 1) | LY2603618 + Desipramine (Period 2) | LY2603618 + Gemcitabine (Continued Access) | LY2603618 + Pemetrexed (Continued Access)
Started | 20 | 0 | 0 | 0
Received at Least 1 Dose of Study Drug | 20 | 0 | 0 | 0
Completed | 20 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Desipramine (Period 1) | LY2603618 + Desipramine (Period 2) | LY2603618 + Gemcitabine (Continued Access) | LY2603618 + Pemetrexed (Continued Access)
Started | 0 | 20 | 0 | 0
Received at Least 1 Dose of Study Drug | 0 | 19 | 0 | 0
Completed | 0 | 19 | 0 | 0
Not Completed | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Period: Continued Access Phase
Arm/Group | Desipramine (Period 1) | LY2603618 + Desipramine (Period 2) | LY2603618 + Gemcitabine (Continued Access) | LY2603618 + Pemetrexed (Continued Access)
Started | 0 | 0 | 12 | 7
Received at Least 1 Dose of Study Drug | 0 | 0 | 12 | 7
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 12 | 7
Not completed — Progression of Disease | 0 | 0 | 8 | 4
Not completed — Protocol Violation | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 0
Not completed — Death | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- All Participants: Single 50-milligram (mg) oral dose of desipramine on Day 1 of Study Period 1. Single 275-mg intravenous infusion over one hour of LY2603618 followed by single 50-mg oral dose of desipramine on Day 1 of Study Period 2.
  Participants may have received additional doses of LY2603618 in combination as follows: 1000 milligrams per square meter (mg/m²) intravenous administration over 30 minutes of gemcitabine on Days 1, 8 and 15 and 230-mg intravenous infusion over one hour of LY2603618 on Days 2, 9 and 16 of 28-day cycles during continued access phase OR 500-mg/m² intravenous administration over 10 minutes of pemetrexed on Day 1 and 275-mg intravenous infusion over one hour of LY2603618 on Day 2 of 21-day cycles during continued access phase.
  Participants were allowed to continue to receive the combination therapy until fulfilling one of the criteria for discontinuation, such as unacceptable toxicity or disease progression.
Arm/Group | All Participants
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 12
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Plasma Pharmacokinetics of LY2603618: the Maximum Concentration of LY2603618 in the Plasma (Cmax)
Time Frame: Period 2 only: Predose, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120 and 144 hours post dose
Population: All participants who received LY2603618 and had pharmacokinetic data collected to calculate the Cmax of LY2603618 in Period 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Groups:
- LY2603618: Single 50-milligram (mg) oral dose of desipramine on Day 1 of Study Period 1.
  Single 275-mg intravenous infusion over one hour of LY2603618 followed by single 50-mg oral dose of desipramine on Day 1 of Study Period 2.
Arm/Group | LY2603618
Number analyzed (Participants) | 19
nanograms/milliliter (ng/mL) | 5950 (39)

2. Primary Outcome: Plasma Pharmacokinetics of Desipramine: the Maximum Concentration of Desipramine in the Plasma (Cmax)
Time Frame: Periods 1 and 2: Predose, 0.5, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 144 and 168 hours post dose
Population: All participants who received desipramine and had pharmacokinetic data collected to calculate the Cmax of desipramine in Periods 1 and 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Groups:
- Desipramine: Single 50-milligram (mg) oral dose of desipramine on Day 1 of Study Period 1.
  Single 275-mg intravenous infusion over one hour of LY2603618 followed by single 50-mg oral dose of desipramine on Day 1 of Study Period 2.
Arm/Group | Desipramine
Number analyzed (Participants) | 20
nanograms/milliliter (ng/mL)
  Period 1 | 21.2 (67)
  Period 2: number analyzed (Participants) | 19
  Period 2 | 22.8 (62)

3. Primary Outcome: Plasma Pharmacokinetics of LY2603618: the Area Under the Plasma Concentration Versus Time Curve From Time Zero to Infinity [AUC(0-∞)]
Time Frame: Period 2 only: Predose, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120 and 144 hours post dose
Population: All participants who received LY2603618 and had pharmacokinetic data collected to calculate the AUC(0-∞) of LY2603618 in Period 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter (ng*h/mL)
Arm/Group | LY2603618
Number analyzed (Participants) | 19
nanograms*hour/milliliter (ng*h/mL) | 53700 (55)

4. Primary Outcome: Plasma Pharmacokinetics of Desipramine: the Area Under the Plasma Concentration Versus Time Curve From Time Zero to Infinity [AUC(0-∞)]
Time Frame: Periods 1 and 2: Predose, 0.5, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 144 and 168 hours post dose
Population: All participants who received desipramine and had pharmacokinetic data collected to calculate the AUC(0-∞) of desipramine in Periods 1 and 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter (ng*h/mL)
Arm/Group | Desipramine
Number analyzed (Participants) | 20
nanograms*hour/milliliter (ng*h/mL)
  Period 1 | 655 (84)
  Period 2: number analyzed (Participants) | 19
  Period 2 | 687 (80)

5. Primary Outcome: Plasma Pharmacokinetics of LY2603618: the Area Under the Plasma Concentration Versus Time Curve From Time Zero to the Last Observed Plasma Concentration of LY2603618 [AUC(0-tlast)]
Time Frame: Period 2 only: Predose 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120 and 144 hours post dose
Population: All participants who received LY2603618 and had pharmacokinetic data collected to calculate the AUC(0-tlast) of LY2603618 in Period 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter (ng*h/mL)
Arm/Group | LY2603618
Number analyzed (Participants) | 19
nanograms*hour/milliliter (ng*h/mL) | 53000 (52)

6. Primary Outcome: Plasma Pharmacokinetics of Desipramine: the Area Under the Plasma Concentration Versus Time Curve From Time Zero to the Last Observed Plasma Concentration of Desipramine [AUC(0-tlast)]
Time Frame: Periods 1 and 2: Predose, 0.5, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 144 and 168 hours post dose
Population: All participants who received desipramine and had pharmacokinetic data collected to calculate AUC(0-tlast) of desipramine in Periods 1 and 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter (ng*h/mL)
Arm/Group | Desipramine
Number analyzed (Participants) | 20
nanogram*hour/milliliter (ng*h/mL)
  Period 1 | 619 (76)
  Period 2: number analyzed (Participants) | 19
  Period 2 | 653 (72)

7. Secondary Outcome: Number of Participants With a Tumor Response
Description: Tumor response is complete response (CR) + partial response (PR), as classified by the investigators according to the Response Evaluation Criteria In Solid Tumors (RECIST) criteria (Version 1.1). CR is the disappearance of all target and non-target lesions and PR is a ≥30% decrease in sum of longest diameter of target lesions. Number of participants with a tumor response is the total number of participants with CR or PR.
Time Frame: Baseline to study completion up to 11 cycles of 21-day cycles
Population: All participants who received at least 1 dose of study drug and had tumor response measured during continued access phase.
Measure: Count of Participants; unit: Participants
Arm/Group | LY2603618 + Gemcitabine (Continued Access) | LY2603618 + Pemetrexed (Continued Access)
Number analyzed (Participants) | 9 | 6
Participants | 1 | 0

ADVERSE EVENTS:
Arm/Group | Desipramine (Period 1) | LY2603618 + Desipramine (Period 2) | LY2603618 + Gemcitabine (Continued Access) | LY2603618 + Pemetrexed (Continued Access)
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/19 | 4/12 | 2/7
Other Adverse Events (participants affected / at risk) | 8/20 | 12/19 | 12/12 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Desipramine (Period 1) (N=20) | LY2603618 + Desipramine (Period 2) (N=19) | LY2603618 + Gemcitabine (Continued Access) (N=12) | LY2603618 + Pemetrexed (Continued Access) (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthritis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Event resulted in death
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Desipramine (Period 1) (N=20) | LY2603618 + Desipramine (Period 2) (N=19) | LY2603618 + Gemcitabine (Continued Access) (N=12) | LY2603618 + Pemetrexed (Continued Access) (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 6 (6) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 8 (11) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 4 (6) | 2 (2)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (6) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 6 (8) | 3 (4)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 5 (6) | 5 (7) | 5 (9)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (4) | 5 (12) | 3 (5)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Disease progression (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2) | 9 (11) | 5 (7)
Injection site reaction (General disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 4 (9) | 1 (1)
Helicobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 4 (4) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 4 (4) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (5) | 2 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema genital (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days